CLINICAL TRIAL: NCT06841913
Title: The Effects of Woodsmoke Exposure on Nasal Immune Responses to Influenza Infection in Normal Human Volunteers
Brief Title: Woodsmoke Exposure, Influenza Infection, and Nasal Immunity
Acronym: SmokeyFlu
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely but potentially may resume
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-1802; 1R01ES036209-01 (NIH)
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Smoke Exposure; Influenza
Keywords: LAIV; Flumist; Influenza; Wood Smoke; Smoke; Fire
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Intervention Model Description: 25% of participants (N=100 total for the study) will undergo each of the following.
  Wood smoke followed by LAIV (N=25) Wood smoke followed by Placebo (N=25) Clean Air followed by LAIV (N=25) Clean Air followed by Placebo (N=25)
  Males and females will be equally enrolled into each of the above cohorts.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a randomized, double-blinded study so packaging and labeling by IDS is such that both study participants and study personnel (lab techs) will be blinded to the treatment (either LAIV or placebo) given. Due to the smell of the WS it will not be possible to completely blind subjects or coordinators as to exposure. The contractor maintaining the woodsmoke exposure chamber add a small amount of woodsmoke into the chamber to minimize bias. The risk for bias is felt to be minimal because all of the study's primary and most of the secondary outcomes are laboratory assays for which the technicians performing the assays will be blinded as to subject group. Unblinding will occur at the conclusion of the study or earlier if needed for safety purposes and as dictated by the UNC IRB, study sponsor, and DSMB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Wood smoke followed by LAIV (Experimental): Participants will receive LAIV after a 2 hour wood smoke exposure.
  Interventions: Biological: LAIV nasal vaccine is chosen as a model viral infection; Other: Wood smoke
- Wood smoke followed by Placebo (Active Comparator): Participants will receive a LAIV placebo after a 2 hour wood smoke exposure.
  Interventions: Other: Wood smoke; Biological: Placebo for LAIV nasal vaccine is chosen as a model viral infection
- Clean Air followed by LAIV (Active Comparator): Participants will receive LAIV after a 2 hour clean air exposure.
  Interventions: Biological: LAIV nasal vaccine is chosen as a model viral infection; Other: Placebo for Wood Smoke (clean Air Exposure)
- Clean Air followed by Placebo (Placebo Comparator): Participants will receive a LAIV placebo after a 2 hour clean air exposure.
  Interventions: Biological: Placebo for LAIV nasal vaccine is chosen as a model viral infection; Other: Placebo for Wood Smoke (clean Air Exposure)

INTERVENTIONS:
Biological: LAIV nasal vaccine is chosen as a model viral infection — Inoculation with LAIV
  Other Names: Live Attenuated Influenza Vaccine; Flumist
  Arms: Clean Air followed by LAIV; Wood smoke followed by LAIV
Other: Wood smoke — Wood smoke exposure concentrations at 500 ug/m3 for two hours.
  Arms: Wood smoke followed by LAIV; Wood smoke followed by Placebo
Biological: Placebo for LAIV nasal vaccine is chosen as a model viral infection — Placebo for LAIV inoculation. Nasal administration of normal saline.
  Arms: Clean Air followed by Placebo; Wood smoke followed by Placebo
Other: Placebo for Wood Smoke (clean Air Exposure) — Clean Air Exposure for 2 hours
  Arms: Clean Air followed by LAIV; Clean Air followed by Placebo

SUMMARY:
This study will investigate the effects of woodsmoke (WS) exposure on human nasal mucosal immune responses to viral infection. The study tests the hypotheses that WS exposure modifies biomarkers of nasal mucosal immune function, increases in Live Attenuated Influenza Virus (LAIV) -induced nasal symptoms, and reduces mucosal antibody production.

DETAILED DESCRIPTION:
This study will investigate the effects of woodsmoke (WS) exposure on human nasal mucosal immune responses to viral infection. The study tests the hypotheses that WS exposure modifies biomarkers of nasal mucosal immune function, increases LAIV-induced nasal symptoms, and reduces mucosal antibody production. Healthy volunteers will be randomized for a 2-hr exposure to WS or placebo (filtered air) and then inoculated with either live attenuated influenza virus (LAIV) or placebo. Nasal mucosal samples, symptoms, and peripheral blood will be collected on days 1,2,3,7, and 21 post-exposure/LAIV and assessed for a) mucosal antiviral responses using targeted and non-targeted analysis of the secretome and tissue-level gene expression; b) symptoms, virus quantity, differential cell count, and virus-specific antibody levels; and c) biomarker signatures associated with infection outcomes using computational modeling tools.

ELIGIBILITY:
Inclusion Criteria:

* Normal lung function,
* oxygen saturation of >94%,
* normal blood pressure,
* no respiratory symptoms on history, no abnormalities on exam, normal pulmonary function testing,
* 18-49 Years of age.

Exclusion Criteria:

* A history of significant chronic illnesses (to include diabetes, autoimmune diseases, immunodeficiency state, known ischemic heart disease, chronic respiratory diseases such as chronic obstructive pulmonary disease or asthma, hypertension)
* Positive pregnancy test within 48 hours of the time of challenge
* Use of any inhaled substance (for medical or recreational purposes).
* Nonsmokers must have been abstinent from smoking for the prior 12 months, having not smoked more than 1 pack over the course of the previous year.
* History of allergy to eggs
* Acute, non-chronic, medical conditions, including (but not limited to) pneumonia or bronchitis requiring antibiotics, febrile illnesses, flu-like symptoms must be totally resolved symptomatically for 3 weeks
* Unspecified illnesses, which in the judgment of the investigator increase the risk associated with the experimental LAIV infection, will be a basis for exclusion.
* Expected exposure of subject to immunocompromised individuals (who can be infected by LAIV) for the 3 weeks following LAIV inoculation.
* Use of immunosuppressive drugs within the past 6 months.
* Previous Woodsmoke exposure <3 weeks, which is considered to an appropriate washout period

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Nasal Mucosal secretome (AUC) | Day 0 to Day 7
  Analysis of the nasal mucosal secretome (secreted factors identified as responsive to WS and/or LAIV). Area under the curve (AUC) will be calculated for each proteomic profile. Descriptive statistics (means and standard deviations) will be computed for outcomes of interest (AUCs), assuming normal distribution as in previous studies.
Gene Expression (AUC) | Day 0 to Day 7
  Tissue-level gene expression (genes identified as responsive to WS and/or LAIV) and assessed for: tissue-level gene expression and untargeted metabolomic and proteomic profiles. Area under the curve (AUC) will be calculated for each gene profile. Descriptive statistics (means and standard deviations) will be computed for outcomes of interest (AUCs), assuming normal distribution as in previous studies.
Virus Quantity (AUC) | Day 0 to Day 7
  Virus quantity in nasal secretions
Nasal Neutrophils (AUC) | Day 0 to Day 7
  nasal secretion
Nasal Viral Antibodies (AUC) | Day 0 to Day 7
  virus-specific antibody levels in nasal secretions
Blood Viral Antibodies (AUC) | Day 0 to Day 7
  virus-specific antibody levels in blood

SECONDARY OUTCOMES:
Peak Tissue gene expression | Day 0 to Day 21
  Peak value of Tissue-level gene expression (genes identified as responsive to WS and/or LAIV)
Peak nasal secretome | Day 0 to Day 21
  Peak Analysis value of the nasal mucosal secretome (secreted factors identified as responsive to WS and/or LAIV)
Peak Nasal Virus quantity | Day 0 to day 21
  Peak value of Virus quantity in nasal secretions
Peak nasal neutrophils | Day 0 to Day 21
  Peak value of nasal neutrophils
Peak Nasal virus anti-bodies | Day 0 to Day 21
  Peak value of virus-specific antibody levels in nasal secretions
Peak blood virus anti-bodies | Day 0 to Day 21
  Peak value of virus-specific antibody levels in blood
Peak Day of Tissue Gene Expression | Day 0 to Day 21
  Peak Day of Tissue-level gene expression (genes identified as responsive to WS and/or LAIV)
Peak Day of nasal secretome | Day 0 to Day 21
  Peak Analysis Day of the nasal mucosal secretome (secreted factors identified as responsive to WS and/or LAIV)
Peak Day of Nasal Virus quantity | Day 0 to day 21
  Peak Day of Virus quantity in nasal secretions
Peak Day of nasal neutrophils | Day 0 to Day 21
  Peak Day of nasal secretion
Peak Day of Nasal virus anti-bodies | Day 0 to Day 21
  Peak day of virus-specific antibody levels in nasal secretions
Peak Day of blood virus anti-bodies | Day 0 to Day 21
  Peak Day of virus-specific antibody levels in blood
Peak Symptom score | Day 0-21
  Flu symptom questionnaire. A score from 0-18 will be recorded. Zero being symptom free and 18 the most symptomatic.
Peak day of symptom score | Day 0-21
  Flu symptom questionnaire. A score from 0-18 will be recorded. Zero being symptom free and 18 the most symptomatic. The day in which there is the highest score will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Rebuli, PhD, Principal Investigator — UNC; Terry Noah, MD, Principal Investigator — UNC
Locations (1):
- Human Studies Facility, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary and Secondary Outcomes data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: The investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
URL: https://guides.lib.unc.edu/nih-data-sharing